CLINICAL TRIAL: NCT06865339
Title: TRIPL: Thoracic Radiotherapy and Inhibition of PD-1 and LAG-3 for Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Thoracic Radiotherapy and Inhibition of PD-1 and LAG-3 for Locally Advanced Non-Small Cell Lung Cancer
Acronym: TRIPL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nitin Ohri (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Henry Ford Health System (Other); NYU Langone Health (Other); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Nitin Ohri, Principal Investigator, Albert Einstein College of Medicine
Organization: Albert Einstein College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-16318
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: NSCLC; Locally Advanced
Keywords: Human Immunoglobulin G (IgG) anti-PD-1 monoclonal antibody; Human IgG anti-lymphocyte activation gene; Tumor Proportion Score
MeSH Terms: interventions — cemiplimab; Radiotherapy

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: PD-L1 (TPS ≥ 50%) (Experimental): * Fixed-dose combination (FDC) of Cemiplimab 350mg IV + Fianlimab 1600mg IV every 3 weeks x 3 cycles
  * Radiotherapy
  * FDC of Cemiplimab + Fianlimab every 3 weeks x 13 cycles, starting 4-6 weeks after completion of RT
  Interventions: Drug: Cemiplimab; Drug: Fianlimab; Radiation: Radiotherapy
- Cohort 2: PD-L1 (TPS < 50%) (Experimental): * FDC of Cemiplimab 350mg IV + Fianlimab 1600mg IV and histology-specific platinum-doublet chemotherapy (PDC) every 3 weeks x 3 cycles
  * Radiotherapy +/- PDC
  * FDC of Cemiplimab + Fianlimab every 3 weeks x 13 cycles, starting 4-6 weeks after completion of RT
  Weekly radiosensitizing PDC will be recommended for PD-L1 TPS <50% patients during RT but is not required
  Interventions: Drug: Cemiplimab; Drug: Fianlimab; Radiation: Radiotherapy; Drug: Platinum Doublet Chemotherapy (PDC)

INTERVENTIONS:
Drug: Cemiplimab — Human IgG anti-PD-1 monoclonal antibody approved for treatment of advanced NSCLC with PD-L1 TPS ≥ 50% as monotherapy and in combination with chemotherapy
  Other Names: REGN2810 (PD1)_cemiplimab_LIBTAYO
Drug: Fianlimab — Human IgG anti-lymphocyte activation gene 3 (LAG-3) monoclonal antibody, which is expressed by various immune cells, and regulates effector T-cell activation and responses. LAG-3 inhibition restores the effector function of exhausted T cells, enhancing their ability to attack tumor cells. Fianlimab is currently under investigation in several clinical studies involving NSCLC (NCT05800015, NCT03916627, NCT05785767).
Radiation: Radiotherapy — Thoracic radiotherapy. Conventionally fractionated 1.8-2.0 Gray (Gy) per day. Adaptive radiotherapy will not be performed unless difficulty with patient setup or changes in internal patient anatomy require repeating the CT simulation procedure
Drug: Platinum Doublet Chemotherapy (PDC) — Acceptable histology-specific PDC regimens include carboplatin plus paclitaxel or nab-paclitaxel (any histology), carboplatin/cisplatin plus pemetrexed (nonsquamous), carboplatin/cisplatin plus etoposide (any histology), and carboplatin/cisplatin plus docetaxel or gemcitabine (squamous). Carboplatin can be used instead of cisplatin after cycle 1 in cases of cisplatin-induced neuro-/oto-/nephrotoxicity as long as the patient remains eligible for chemoradiotherapy. Weekly radiosensitizing PDC will be recommended for PD-L1 TPS <50% patients during RT but is not required.
  Arms: Cohort 2: PD-L1 (TPS < 50%)

SUMMARY:
Determine anti-tumor efficacy by characterizing response rates on positron emission tomography (PET) following three cycles of induction immunotherapy with cemiplimab and fianlimab without chemotherapy for locally advanced non-small cell lung cancer (LA-NSCLC).

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) represents more than 80% of lung cancers, and approximately 35% of NSCLC patients present with stage III disease. Standard treatment for patients with locally advanced NSCLC, which may be defined as American Joint Committee on Cancer (AJCC) stage III disease or unresectable stage II disease, typically consists of conventionally fractionated (1.8-2.0 Gray (Gy) per day) radiotherapy (RT) to a total dose of approximately 60 Gy with concurrent chemotherapy. Based on the PACIFIC trial (NCT02125461), patients without disease progression after concurrent chemoradiotherapy are typically offered a one-year course of the adjuvant PD-L1 inhibitor durvalumab, regardless of PD-L1 tumor proportion score (TPS). Recent results from the PACIFIC-2 trial (NCT03519971) failed to demonstrate a survival benefit of adding concurrent durvalumab to chemoradiotherapy, and therefore the PACIFIC regimen of adjuvant immunotherapy following chemoradiation remains the standard of care for unresectable LA-NSCLC.

Based on the PACIFIC trial standard, both the RT and systemic therapy utilized to treat LA-NSCLC patients in standard of care follow a non-biomarker selected "one-size-fits-all" approach in the US. In advanced NSCLC, however, patients with high PD-L1 TPS score (≥ 50%) benefit more from the immune checkpoint inhibitors pembrolizumab, atezolizumab, and cemiplimab compared to cytotoxic chemotherapy alone, and single agent immunotherapy (IO) has become a first-line standard of care for such patients. Omitting chemotherapy from the treatment of LA-NSCLC patients with high PD-L1 expression who will receive IO is a logical step. On the other hand, patients with low PD-L1 TPS score (< 50%) benefit less from single agent IO in advanced NSCLC, and IO is typically offered together with chemotherapy. Given the poor response to IO for patients with low PD-L1 TPS expression, the investigator team believes that combination IO plus chemotherapy could be particularly beneficial in the low-TPS LA-NSCLC setting.

Induction (also referred to as neoadjuvant) IO before RT for LA-NSCLC has several potential advantages. For example, the native tumor functioning as an in-situ vaccine in the neoadjuvant setting, with an intact lymphatic system and unirradiated nodal status, could promote optimal immune priming. Indeed, neoadjuvant IO has shown impressive efficacy in both deficient mismatch repair (dMMR) rectal cancer and melanoma. For early-stage NSCLC, this approach is highlighted in recent neoadjuvant trials of immune checkpoint inhibition in combination with chemotherapy for resectable NSCLC, such as CheckMate 816 (NCT02998528), Keynote-671 (NCT03425643), and NADIMII (NCT03838159). Furthermore, results from the PACIFIC trial and real-world data show that approximately 25% of LA-NSCLC patients started on chemoradiotherapy never receive consolidation durvalumab, and approximately 50% of patients started on consolidation durvalumab do not complete the intended year of treatment. Thus, administering induction IO may be particularly advantageous for LA-NSCLC patients to enhance IO treatment delivery.

SPRINT (NCT03523702) was a multi-institutional Phase II trial where biomarker-selected (PD-L1 TPS ≥ 50%) LA-NSCLC patients were treated with 3 cycles of induction pembrolizumab to reduce the extent of thoracic RT, and cytotoxic chemotherapy was omitted from the treatment regimen. Patients with PD-L1 TPS < 50% received standard concurrent chemoradiotherapy (chemoRT) followed by standard adjuvant treatment, to serve as a non-randomized comparator for evaluating toxicities and clinical outcomes. Following induction, PD-L1 TPS ≥ 50% patients received PET-based dose-painted RT according to a novel and personalized approach that was studied in two prior trials (NCT02073968, NCT03481114) that can decrease toxicities by utilizing shortened courses of RT and reducing doses administered to small tumors and nodes. Based on these studies, PET response to induction IO using PERCIST criteria may serve as a useful prognostic factor to identify LA-NSCLC patients more likely to respond to novel IO regimens at an earlier time point in treatment (prior to administration of RT). This observation is also supported by prior prospective and retrospective studies showing that response on PET rather than CT may be a better predictor of survival for NSCLC patients receiving IO. Furthermore, early identification of IO response provides added insight to a tumor's unique immune biology that could be used to individualize subsequent RT, IO, and/or chemotherapy treatment plans. Overall, SPRINT demonstrated high treatment efficacy with limited toxicity and introduces PET response to induction IO as a novel endpoint that allows for early assessment of treatment activity, and which could potentially serve as a new paradigm in LA-NSCLC interventional studies.

Based on this experience, the investigator team believes that the SPRINT treatment approach (induction IO followed by RT and consolidation IO) can be used to investigate other novel IO combinations for biomarker-selected LA-NSCLC. One such immune target is lymphocyte activation gene 3 (LAG3), which is expressed by various immune cells, and regulates effector T-cell activation and responses. LAG-3 inhibition restores the effector function of exhausted T cells, enhancing their ability to attack tumor cells. In addition, LAG-3's inhibitory effects on T cells appear distinct from those of PD-L1, serving as a potential rationale for combining LAG-3 and PD-1/PD-L1 inhibition. In metastatic melanoma, the RELATIVITY-047 trial (NCT03470922) showed that combination PD-1 and LAG-3 blockade with nivolumab and relatlimab, respectively, improves progression-free survival (PFS) compared to nivolumab alone with a favorable toxicity versus nivolumab plus the CTLA-4 inhibitor ipilimumab. These findings suggest that combination PD-1 and LAG-3 inhibition may have potential utility for treatment of other malignancies, such as NSCLC. Furthermore, a Phase I study of cemiplimab and fianlimab in unresectable stage IIIB-C or IV NSCLC (NCT03005782) showed that the combination demonstrated clinical activity with a similar safety profile compared to cemiplimab alone. Given the promising findings observed in SPRINT, RELATIVITY-047, and NCT03005782, the research team believes that dual immune checkpoint blockade with the PD-1 inhibitor cemiplimab plus the LAG-3 inhibitor fianlimab administered before and after thoracic RT, as per the SPRINT approach, has valuable therapeutic potential for LA-NSCLC patients.

Treatment will be administered in three phases as detailed in this registration: (1) three cycles of induction IO, with histology-specific platinum doublet chemotherapy (PDC) added for subjects with PD-L1 TPS <50%; (2) thoracic RT (with concurrent PDC recommended for subjects with PD-L1 TPS <50%); (3) 13 cycles of consolidation IO.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated and biopsy-proven NSCLC, with measurable disease (at least 1 unidimensional, radiographically measurable lesion based on RECIST v1.1) and one of the following stages: (prior resection or stereotactic radiotherapy for early-stage disease is allowed)

  * AJCC version 8 Stage II disease, medically or technically unresectable
  * AJCC version 8 Stage III disease, eligible for non-surgical treatment
* Determination of PD-L1 expression on pretreatment tumor specimen using a clinically validated assay
* Eligible for standard nonsurgical treatment for Stage III NSCLC, i.e., chemotherapy and concurrent RT followed by adjuvant durvalumab
* Whole body PET/CT within 42 days prior to study entry demonstrating hypermetabolic pulmonary lesion(s) and/or thoracic lymph node(s)
* MRI of the brain or head CT with contrast within 42 days prior to study entry
* PFTs within 42 days of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate end-organ function for study therapy, as per clinician assessment and including:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
  * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
  * AST (SGOT)/ALT (SGPT), and alkaline phosphatase ≤ 2.5 x institutional upper limit of normal (ULN)
  * Serum creatinine clearance >30 mL/min by the Cockcroft-Gault formula (as below) or by 24-hour urine collection for determination of creatinine clearance: (except for patients planned to receive pemetrexed, in which case serum creatinine clearance needs to >45 ml/min)

    * Males: Weight (kg) x (140 - Age) ÷ (72 x serum creatinine (mg/dL))
    * Females: 0.85 x Weight (kg) x (140 - Age) ÷ (72 x serum creatinine (mg/dL))
* A female participant is eligible to participate if she is not pregnant (see Exclusion Criteria), not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) as defined in the Appendix
  * A WOCBP who agrees to follow the contraceptive guidance in the Appendix during the treatment period and for at least 6 months (180 days) after the last dose of study treatment with cemiplimab and fianlimab
  * A WOCBP who agrees to follow the contraceptive guidance in the Appendix and for at least 6 months after the last dose of chemotherapy or as specified in FDA prescribing labels (e.g. 14 months after the last dose of cisplatin)
* A male participant must agree to use contraception during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial

Exclusion Criteria:

* Presence of known sensitizing epidermal growth factor (EGFR) mutation or anaplastic lymphoma kinase (ALK) fusion

  o Determination of EGFR/ALK mutation status is required for non-squamous cell carcinoma histologies and recommended for squamous cell carcinoma
* Prior therapy with an anti-PD-1, anti-PD-L1, or LAG-3 inhibitor
* Patient currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Active malignancy other than lung cancer that (1) requires active treatment other than hormonal therapy and (2) is deemed by the treating physicians to be likely to affect the patient's life expectancy
* A history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Known history of myocarditis
* Troponin T (TnT) or troponin I (TnI) > 2x institutional ULN at baseline. Patients with TnT or TnI levels between > 1 to 2x ULN are permitted if repeat levels within 24 hours are ≤ 1x ULN. If TnT or TnI levels are > 1 to 2x ULN within 24 hours, the subject may undergo a cardiac evaluation and be considered for treatment by the investigator based on the medical judgement in the patient's best interest
* Known active Bacillus Tuberculosis (TB)
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnancy, assessed with urine pregnancy test within 72 hours prior to study treatment allocation. If urine pregnancy test is positive or cannot be confirmed as negative, a serum pregnancy test is required. If more than 72 hours elapse between screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative
* Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment
* History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (e.g., cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication
* Active infection requiring therapy
* Uncontrolled infection with HIV, Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection

  * Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards
  * Patients with known hepatitis B (HepBsAg+) who have controlled infection (serum hepatitis B virus DNA PCR that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards and must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study drug
  * Patients who are known hepatitis C virus antibody positive (HCV Ab+) who have controlled infection (undetectable HCV RNA by polymerase chain reaction (PCR) either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted
  * Patients with HIV or hepatitis must be reviewed by a qualified specialist (e.g., infectious disease or hepatologist) managing this disease prior to commencing and regularly throughout the duration of their participation in the trial
* Diagnosis of immunodeficiency or ongoing chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Known hypersensitivity to the active substances or to any of the excipients
* Received a live vaccine within 30 days of planned start of study medication o Live or live attenuated vaccination with replicating potential. If a patient intends to receive a COVID-19 vaccine before the start of study drug, participation in the study should be delayed at least 1 week after any COVID-19 vaccination. During the treatment period, it is recommended to delay COVID-19 vaccination until patients are receiving and tolerating a steady dose of study drug. A vaccine dose should not be less than 48 hours before or after study drug dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) to induction IO therapy | Following 3 cycles (each cycle is ~3 weeks) of induction IO therapy, approximately 10 weeks overall
  ORR to induction therapy will be evaluated by fluorodeoxyglucose (FDG) FDG-PET scan using Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) criteria. Pre-and post-treatment maximum standardized uptake value (SUV) levels following PERCIST criteria will be assessed. Specifically, the percentage of patients who experience either a complete metabolic response (CMR) or partial metabolic response (PMR) based on changes in FDG uptake will be determined and quantified using the following calculation (PMR+CMR/Sample Size). All participants who initiate study therapy will be analyzed for ORR. Participants who do not undergo response rate evaluation for any reason will be categorized as non-responders. Response rates in each study cohort will be summarized and reported using counts and percentages. 95% Clopper-Pearson confidence intervals will be calculated. ORR based on PET are more accurate predictors of long-term clinical outcomes than computed tomography (CT).

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) | From initiation of study immunotherapy until 4 weeks following completion of radiotherapy, up to 17 weeks total
  DLT will be defined as the occurrence of any of the following adverse events (AEs) that, in the opinion of the PI, significantly interferes with the patient's optimal management:
  * CTCAE v5.0 Grade 3-4 or recurrent grade 2 pneumonitis; Grade 4 diarrhea/colitis; Grade 3-4 myocarditis; or Grade 3 thrombocytopenia with clinically significant bleeding
  * Febrile neutropenia (any grade)
  * Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥3 times upper limit of normal (ULN) with concurrent increase in total bilirubin >2 times ULN, without evidence of cholestasis or alternative explanations such as viral hepatitis, disease progression in the liver, etc. (i.e., Hy's Law).
  * any death not clearly due to the underlying disease or extraneous causes
  * any toxicity requiring permanent discontinuation of study drug(s).
  DLTs will be assessed as a dichotomous (Yes/No) measure. Results will be summarized and reported by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Ohri, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Einstein Comprehensive Cancer Center (MECCC), The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi AP, Tang XY, Xiong YL, Zheng KF, Liu YJ, Shi XG, Lv Y, Jiang T, Ma N, Zhao JB. Immune Checkpoint LAG3 and Its Ligand FGL1 in Cancer. Front Immunol. 2022 Jan 17;12:785091. doi: 10.3389/fimmu.2021.785091. eCollection 2021. PMID 35111155
- [Background] Peters S CB, Luft A, et al: Association between KRAS/STK11/KEAP1 mutations and outcomes in POSEIDON: Durvalumab ± tremelimumab + chemotherapy in mNSCLC. 2022 World Conference on Lung Cancer. Abstract OA15.04., 2022
- [Background] Gartrell RD, Marks DK, Hart TD, Li G, Davari DR, Wu A, Blake Z, Lu Y, Askin KN, Monod A, Esancy CL, Stack EC, Jia DT, Armenta PM, Fu Y, Izaki D, Taback B, Rabadan R, Kaufman HL, Drake CG, Horst BA, Saenger YM. Quantitative Analysis of Immune Infiltrates in Primary Melanoma. Cancer Immunol Res. 2018 Apr;6(4):481-493. doi: 10.1158/2326-6066.CIR-17-0360. Epub 2018 Feb 21. PMID 29467127
- [Background] Gartrell-Corrado RD, Chen AX, Rizk EM, Marks DK, Bogardus MH, Hart TD, Silverman AM, Bayan CY, Finkel GG, Barker LW, Komatsubara KM, Carvajal RD, Horst BA, Chang R, Monod A, Rabadan R, Saenger YM. Linking Transcriptomic and Imaging Data Defines Features of a Favorable Tumor Immune Microenvironment and Identifies a Combination Biomarker for Primary Melanoma. Cancer Res. 2020 Mar 1;80(5):1078-1087. doi: 10.1158/0008-5472.CAN-19-2039. Epub 2020 Jan 16. PMID 31948941
- [Background] Gartrell RD, Marks DK, Rizk EM, Bogardus M, Gerard CL, Barker LW, Fu Y, Esancy CL, Li G, Ji J, Rui S, Ernstoff MS, Taback B, Pabla S, Chang R, Lee SJ, Krolewski JJ, Morrison C, Horst BA, Saenger YM. Validation of Melanoma Immune Profile (MIP), a Prognostic Immune Gene Prediction Score for Stage II-III Melanoma. Clin Cancer Res. 2019 Apr 15;25(8):2494-2502. doi: 10.1158/1078-0432.CCR-18-2847. Epub 2019 Jan 15. PMID 30647081
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Spigel DR, Faivre-Finn C, Gray JE, Vicente D, Planchard D, Paz-Ares L, Vansteenkiste JF, Garassino MC, Hui R, Quantin X, Rimner A, Wu YL, Ozguroglu M, Lee KH, Kato T, de Wit M, Kurata T, Reck M, Cho BC, Senan S, Naidoo J, Mann H, Newton M, Thiyagarajah P, Antonia SJ. Five-Year Survival Outcomes From the PACIFIC Trial: Durvalumab After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Apr 20;40(12):1301-1311. doi: 10.1200/JCO.21.01308. Epub 2022 Feb 2. PMID 35108059
- [Background] Bradley J, Sugawara S, Lee KHH, et al: Durvalumab in combination with chemoradiotherapy for patients with unresectable stage III NSCLC: Final results from PACIFIC 2, European Lung Cancer Conference 2024, Annals of Oncology, 2024, pp 1-12
- [Background] Gogishvili M, Melkadze T, Makharadze T, Giorgadze D, Dvorkin M, Penkov K, Laktionov K, Nemsadze G, Nechaeva M, Rozhkova I, Kalinka E, Gessner C, Moreno-Jaime B, Passalacqua R, Li S, McGuire K, Kaul M, Paccaly A, Quek RGW, Gao B, Seebach F, Weinreich DM, Yancopoulos GD, Lowy I, Gullo G, Rietschel P. Cemiplimab plus chemotherapy versus chemotherapy alone in non-small cell lung cancer: a randomized, controlled, double-blind phase 3 trial. Nat Med. 2022 Nov;28(11):2374-2380. doi: 10.1038/s41591-022-01977-y. Epub 2022 Aug 25. PMID 36008722
- [Background] Sezer A, Kilickap S, Gumus M, Bondarenko I, Ozguroglu M, Gogishvili M, Turk HM, Cicin I, Bentsion D, Gladkov O, Clingan P, Sriuranpong V, Rizvi N, Gao B, Li S, Lee S, McGuire K, Chen CI, Makharadze T, Paydas S, Nechaeva M, Seebach F, Weinreich DM, Yancopoulos GD, Gullo G, Lowy I, Rietschel P. Cemiplimab monotherapy for first-line treatment of advanced non-small-cell lung cancer with PD-L1 of at least 50%: a multicentre, open-label, global, phase 3, randomised, controlled trial. Lancet. 2021 Feb 13;397(10274):592-604. doi: 10.1016/S0140-6736(21)00228-2. PMID 33581821
- [Background] Kisielow M, Kisielow J, Capoferri-Sollami G, Karjalainen K. Expression of lymphocyte activation gene 3 (LAG-3) on B cells is induced by T cells. Eur J Immunol. 2005 Jul;35(7):2081-8. doi: 10.1002/eji.200526090. PMID 15971272
- [Background] Grosso JF, Goldberg MV, Getnet D, Bruno TC, Yen HR, Pyle KJ, Hipkiss E, Vignali DA, Pardoll DM, Drake CG. Functionally distinct LAG-3 and PD-1 subsets on activated and chronically stimulated CD8 T cells. J Immunol. 2009 Jun 1;182(11):6659-69. doi: 10.4049/jimmunol.0804211. PMID 19454660
- [Background] Hamid O, Lewis KD, Weise A, McKean M, Papadopoulos KP, Crown J, Kim TM, Lee DH, Thomas SS, Mehnert J, Kaczmar J, Lakhani NJ, Kim KB, Middleton MR, Rabinowits G, Spira AI, Yushak M, Mehmi I, Fang F, Chen S, Mani J, Jankovic V, Wang F, Fiaschi N, Brennan L, Paccaly A, Masinde S, Salvati M, Fury MG, Kroog G, Lowy I, Gullo G. Phase I Study of Fianlimab, a Human Lymphocyte Activation Gene-3 (LAG-3) Monoclonal Antibody, in Combination With Cemiplimab in Advanced Melanoma. J Clin Oncol. 2024 Aug 20;42(24):2928-2938. doi: 10.1200/JCO.23.02172. Epub 2024 Jun 20. PMID 38900987
- [Background] National Comprehensive Cancer Center Network. Non-Small Cell Lung Cancer. (Version 3.2024).
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leal TA, Riess JW, Jensen E, Zhao B, Pietanza MC, Brahmer JR. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50. J Clin Oncol. 2021 Jul 20;39(21):2339-2349. doi: 10.1200/JCO.21.00174. Epub 2021 Apr 19. PMID 33872070
- [Background] Herbst RS, Giaccone G, de Marinis F, Reinmuth N, Vergnenegre A, Barrios CH, Morise M, Felip E, Andric Z, Geater S, Ozguroglu M, Zou W, Sandler A, Enquist I, Komatsubara K, Deng Y, Kuriki H, Wen X, McCleland M, Mocci S, Jassem J, Spigel DR. Atezolizumab for First-Line Treatment of PD-L1-Selected Patients with NSCLC. N Engl J Med. 2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. PMID 32997907
- [Background] Cercek A, Lumish M, Sinopoli J, Weiss J, Shia J, Lamendola-Essel M, El Dika IH, Segal N, Shcherba M, Sugarman R, Stadler Z, Yaeger R, Smith JJ, Rousseau B, Argiles G, Patel M, Desai A, Saltz LB, Widmar M, Iyer K, Zhang J, Gianino N, Crane C, Romesser PB, Pappou EP, Paty P, Garcia-Aguilar J, Gonen M, Gollub M, Weiser MR, Schalper KA, Diaz LA Jr. PD-1 Blockade in Mismatch Repair-Deficient, Locally Advanced Rectal Cancer. N Engl J Med. 2022 Jun 23;386(25):2363-2376. doi: 10.1056/NEJMoa2201445. Epub 2022 Jun 5. PMID 35660797
- [Background] Patel SP, Othus M, Chen Y, Wright GP Jr, Yost KJ, Hyngstrom JR, Hu-Lieskovan S, Lao CD, Fecher LA, Truong TG, Eisenstein JL, Chandra S, Sosman JA, Kendra KL, Wu RC, Devoe CE, Deutsch GB, Hegde A, Khalil M, Mangla A, Reese AM, Ross MI, Poklepovic AS, Phan GQ, Onitilo AA, Yasar DG, Powers BC, Doolittle GC, In GK, Kokot N, Gibney GT, Atkins MB, Shaheen M, Warneke JA, Ikeguchi A, Najera JE, Chmielowski B, Crompton JG, Floyd JD, Hsueh E, Margolin KA, Chow WA, Grossmann KF, Dietrich E, Prieto VG, Lowe MC, Buchbinder EI, Kirkwood JM, Korde L, Moon J, Sharon E, Sondak VK, Ribas A. Neoadjuvant-Adjuvant or Adjuvant-Only Pembrolizumab in Advanced Melanoma. N Engl J Med. 2023 Mar 2;388(9):813-823. doi: 10.1056/NEJMoa2211437. PMID 36856617
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841
- [Background] Wakelee H, Liberman M, Kato T, Tsuboi M, Lee SH, Gao S, Chen KN, Dooms C, Majem M, Eigendorff E, Martinengo GL, Bylicki O, Rodriguez-Abreu D, Chaft JE, Novello S, Yang J, Keller SM, Samkari A, Spicer JD; KEYNOTE-671 Investigators. Perioperative Pembrolizumab for Early-Stage Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):491-503. doi: 10.1056/NEJMoa2302983. Epub 2023 Jun 3. PMID 37272513
- [Background] Provencio M, Nadal E, Gonzalez-Larriba JL, Martinez-Marti A, Bernabe R, Bosch-Barrera J, Casal-Rubio J, Calvo V, Insa A, Ponce S, Reguart N, de Castro J, Mosquera J, Cobo M, Aguilar A, Lopez Vivanco G, Camps C, Lopez-Castro R, Moran T, Barneto I, Rodriguez-Abreu D, Serna-Blasco R, Benitez R, Aguado de la Rosa C, Palmero R, Hernando-Trancho F, Martin-Lopez J, Cruz-Bermudez A, Massuti B, Romero A. Perioperative Nivolumab and Chemotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Aug 10;389(6):504-513. doi: 10.1056/NEJMoa2215530. Epub 2023 Jun 28. PMID 37379158
- [Background] Girard N, Bar J, Garrido P, Garassino MC, McDonald F, Mornex F, Filippi AR, Smit HJM, Peters S, Field JK, Christoph DC, Sibille A, Fietkau R, Haakensen VD, Chouaid C, Markman B, Hiltermann TJN, Taus A, Sawyer W, Allen A, Chander P, Licour M, Solomon B. Treatment Characteristics and Real-World Progression-Free Survival in Patients With Unresectable Stage III NSCLC Who Received Durvalumab After Chemoradiotherapy: Findings From the PACIFIC-R Study. J Thorac Oncol. 2023 Feb;18(2):181-193. doi: 10.1016/j.jtho.2022.10.003. Epub 2022 Oct 25. PMID 36307040
- [Background] Pennock M, Halmos B, Bodner W, Cheng H, Gucalp R, Ohri N. Exploring causes and consequences of early discontinuation of durvalumab after chemoradiotherapy for non-small cell lung cancer. Clin Transl Radiat Oncol. 2023 Jun 1;41:100643. doi: 10.1016/j.ctro.2023.100643. eCollection 2023 Jul. PMID 37346274
- [Background] Ohri N, Jolly S, Cooper BT, Kabarriti R, Bodner WR, Klein J, Guha C, Viswanathan S, Shum E, Sabari JK, Cheng H, Gucalp RA, Castellucci E, Qin A, Gadgeel SM, Halmos B. Selective Personalized RadioImmunotherapy for Locally Advanced Non-Small-Cell Lung Cancer Trial (SPRINT). J Clin Oncol. 2024 Feb 10;42(5):562-570. doi: 10.1200/JCO.23.00627. Epub 2023 Nov 21. PMID 37988638
- [Background] Kaira K, Higuchi T, Naruse I, Arisaka Y, Tokue A, Altan B, Suda S, Mogi A, Shimizu K, Sunaga N, Hisada T, Kitano S, Obinata H, Yokobori T, Mori K, Nishiyama M, Tsushima Y, Asao T. Metabolic activity by 18F-FDG-PET/CT is predictive of early response after nivolumab in previously treated NSCLC. Eur J Nucl Med Mol Imaging. 2018 Jan;45(1):56-66. doi: 10.1007/s00259-017-3806-1. Epub 2017 Aug 21. PMID 28828507
- [Background] Rossi G, Bauckneht M, Genova C, Rijavec E, Biello F, Mennella S, Dal Bello MG, Cittadini G, Bruzzi P, Piva R, Ceriani V, Sambuceti G, Lopci E, Morbelli S, Grossi F. Comparison Between 18F-FDG PET-Based and CT-Based Criteria in Non-Small Cell Lung Cancer Patients Treated with Nivolumab. J Nucl Med. 2020 Jul;61(7):990-998. doi: 10.2967/jnumed.119.233056. Epub 2019 Dec 5. PMID 31806768
- [Background] Andrews LP, Cillo AR, Karapetyan L, Kirkwood JM, Workman CJ, Vignali DAA. Molecular Pathways and Mechanisms of LAG3 in Cancer Therapy. Clin Cancer Res. 2022 Dec 1;28(23):5030-5039. doi: 10.1158/1078-0432.CCR-21-2390. PMID 35579997
- [Background] Tawbi HA, Schadendorf D, Lipson EJ, Ascierto PA, Matamala L, Castillo Gutierrez E, Rutkowski P, Gogas HJ, Lao CD, De Menezes JJ, Dalle S, Arance A, Grob JJ, Srivastava S, Abaskharoun M, Hamilton M, Keidel S, Simonsen KL, Sobiesk AM, Li B, Hodi FS, Long GV; RELATIVITY-047 Investigators. Relatlimab and Nivolumab versus Nivolumab in Untreated Advanced Melanoma. N Engl J Med. 2022 Jan 6;386(1):24-34. doi: 10.1056/NEJMoa2109970. PMID 34986285
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hogg D, Hill A, Marquez-Rodas I, Haanen J, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bastholt L, Rizzo JI, Balogh A, Moshyk A, Hodi FS, Wolchok JD. Five-Year Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2019 Oct 17;381(16):1535-1546. doi: 10.1056/NEJMoa1910836. Epub 2019 Sep 28. PMID 31562797
- [Background] Cascone T, William WN Jr, Weissferdt A, Leung CH, Lin HY, Pataer A, Godoy MCB, Carter BW, Federico L, Reuben A, Khan MAW, Dejima H, Francisco-Cruz A, Parra ER, Solis LM, Fujimoto J, Tran HT, Kalhor N, Fossella FV, Mott FE, Tsao AS, Blumenschein G Jr, Le X, Zhang J, Skoulidis F, Kurie JM, Altan M, Lu C, Glisson BS, Byers LA, Elamin YY, Mehran RJ, Rice DC, Walsh GL, Hofstetter WL, Roth JA, Antonoff MB, Kadara H, Haymaker C, Bernatchez C, Ajami NJ, Jenq RR, Sharma P, Allison JP, Futreal A, Wargo JA, Wistuba II, Swisher SG, Lee JJ, Gibbons DL, Vaporciyan AA, Heymach JV, Sepesi B. Neoadjuvant nivolumab or nivolumab plus ipilimumab in operable non-small cell lung cancer: the phase 2 randomized NEOSTAR trial. Nat Med. 2021 Mar;27(3):504-514. doi: 10.1038/s41591-020-01224-2. Epub 2021 Feb 18. PMID 33603241
- [Background] Gartrell RD, Enzler T, Kim PS, Fullerton BT, Fazlollahi L, Chen AX, Minns HE, Perni S, Weisberg SP, Rizk EM, Wang S, Oh EJ, Guo XV, Chiuzan C, Manji GA, Bates SE, Chabot J, Schrope B, Kluger M, Emond J, Rabadan R, Farber D, Remotti HE, Horowitz DP, Saenger YM. Neoadjuvant chemoradiation alters the immune microenvironment in pancreatic ductal adenocarcinoma. Oncoimmunology. 2022 May 5;11(1):2066767. doi: 10.1080/2162402X.2022.2066767. eCollection 2022. PMID 35558160
- [Background] Casarrubios M, Provencio M, Nadal E, Insa A, Del Rosario Garcia-Campelo M, Lazaro-Quintela M, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe R, Vinolas N, Barneto Aranda I, Massuti B, Sierra-Rodero B, Martinez-Toledo C, Fernandez-Miranda I, Serna-Blanco R, Romero A, Calvo V, Cruz-Bermudez A. Tumor microenvironment gene expression profiles associated to complete pathological response and disease progression in resectable NSCLC patients treated with neoadjuvant chemoimmunotherapy. J Immunother Cancer. 2022 Sep;10(9):e005320. doi: 10.1136/jitc-2022-005320. PMID 36171009
- [Background] Laza-Briviesca R, Cruz-Bermudez A, Nadal E, Insa A, Garcia-Campelo MDR, Huidobro G, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Massuti B, Casarrubios M, Sierra-Rodero B, Tarin C, Garcia-Grande A, Haymaker C, Wistuba II, Romero A, Franco F, Provencio M. Blood biomarkers associated to complete pathological response on NSCLC patients treated with neoadjuvant chemoimmunotherapy included in NADIM clinical trial. Clin Transl Med. 2021 Jul;11(7):e491. doi: 10.1002/ctm2.491. PMID 34323406
- [Background] Langendijk H, Aaronson NK, de Jong JM, ten Velde GP, Muller MJ, Wouters M. The prognostic impact of quality of life assessed with the EORTC QLQ-C30 in inoperable non-small cell lung carcinoma treated with radiotherapy. Radiother Oncol. 2000 Apr;55(1):19-25. doi: 10.1016/s0167-8140(00)00158-4. PMID 10788684
- [Background] Fayers P, Bottomley A; EORTC Quality of Life Group; Quality of Life Unit. Quality of life research within the EORTC-the EORTC QLQ-C30. European Organisation for Research and Treatment of Cancer. Eur J Cancer. 2002 Mar;38 Suppl 4:S125-33. doi: 10.1016/s0959-8049(01)00448-8. PMID 11858978
- [Background] Werner-Wasik M, Nelson AD, Choi W, Arai Y, Faulhaber PF, Kang P, Almeida FD, Xiao Y, Ohri N, Brockway KD, Piper JW, Nelson AS. What is the best way to contour lung tumors on PET scans? Multiobserver validation of a gradient-based method using a NSCLC digital PET phantom. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):1164-71. doi: 10.1016/j.ijrobp.2010.12.055. Epub 2011 Apr 29. PMID 21531085
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774